CLINICAL TRIAL: NCT06635694
Title: naVIGation Invitations Liver surveillANce upTake
Acronym: VIGILANT
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: RM Partners (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23HH8630
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Chronic Hep B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Responsible clinician will request surveillance imaging and ultrasound appointment will be booked using an automated call/recall system. A formal invitation to surveillance and an informational sheet will be sent by post to patient's home address, addressing concerns including fear, and FAQs e.g. duration of scan and level of discomfort. Patients will receive a reminder 2 weeks prior to their appointment. Results will be automatically sent to the relevant hepatology unit and GP. Patients will be informed of results by mail or through "patientknowsbest" app, and invited for repeat ultrasound in 6 months. Patients with abnormal results will be contacted by the direct care team to organise further investigations. Non-attendance will be followed by a further appointment letter/text. Patients who fail to attend 2 appointments will be contacted by the direct care team. Their reasons for non-attendance will be recorded and GP contacted.
- Patient Navigator: Patients will receive usual care plus a scripted phone call from a Patient Navigator the week prior to the surveillance appointment to remind patients, offer to reschedule the appointment if the patient is unable to attend, and address any concerns about the appointment. All other procedures will be the same as usual care. Additionally, Navigators will call patients who have not attended surveillance imaging appointments to explore any barriers to attendance and how these might be addressed.

SUMMARY:
This study aims to evaluate the efficacy of Patient Navigators and mailed surveillance invitations on attendance of Hepatocellular Carcinoma (HCC) ultrasound surveillance appointments. The investigators hypothesise that mailed invitations and Patient Navigators will improve attendance at HCC surveillance appointments and increase the proportion of patients diagnosed at an early stage, compared with a control group receiving usual care.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer-related death worldwide. Despite advances in treatment options, prognosis remains worrying, with 5-year survival rates remaining less than 20%.

Surveillance for HCC involves six-monthly ultrasounds (US) of the liver and has been demonstrated to increase rate of early diagnosis, which translates to improved survival. However, the uptake of HCC surveillance is low internationally; in Western countries, only 20% of patients eligible for HCC surveillance receive a surveillance test.

The current provision of HCC surveillance in the UK is ad hoc: eligible patients have six-monthly ultrasound requested by their clinician (usually a gastroenterologist, hepatologist or hepatology clinical nurse specialist). Patients receive an ultrasound appointment in the post with no formal invitation or information about the surveillance test. Work with focus groups suggests lack of knowledge and fear are barriers to HCC surveillance attendance.

Previous research has shown that patient navigation increased HCC surveillance uptake in an American population. However, there has been no research on interventions aimed at improving surveillance uptake in the UK population.

The study predicts that the mailed invitations and Patient Navigators will improve patient attendance at HCC surveillance and increases the number of patients diagnosed with early-stage HCC, compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ECOG performance status of 0-2
* Eligible for HCC surveillance as defined by NICE and EASL criteria
* Child Pugh A or B cirrhosis
* Child Pugh C cirrhosis AND on liver transplant waiting list
* High risk chronic hepatitis B

Exclusion Criteria:

* Previous or current diagnosis of HCC
* Child Pugh C cirrhosis
* Frailty (Clinical Frailty Scale >7)
* Previous liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving 6-monthly ultrasound surveillance for HCC
Sampling Method: Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-08-19 (Estimated); Study Completion 2027-08-19 (Estimated)

PRIMARY OUTCOMES:
Attendance rates at 6-months intervals | 2 years
Proportion of patients in each arm attending HCC surveillance regularly | 2 years

SECONDARY OUTCOMES:
Proportion of patients in each arm diagnosed with HCC compared with late-stage HCC | 2 years
Cost of intervention compared to standard of care | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pandiaraja M, Qurashi M, Izadi H, Martinez M, Sharma R. Efficacy of mailed surveillance invitations and telephone patient navigation to improve hepatocellular carcinoma surveillance uptake: study protocol of VIGILANT-a single-centre, two-arm randomised controlled trial. BMJ Open. 2025 Jun 30;15(6):e097162. doi: 10.1136/bmjopen-2024-097162. PMID 40588390